CLINICAL TRIAL: NCT04691726
Title: Randomized, Double-blind, Placebo-controlled Single-centre Clinical Trial Evaluating Efficacy and Safety of Intraoperative and Postoperative Continuous Lidocaine Infusion in High Cardiac Risk Vascular Surgery
Brief Title: Impact of Intra- and Postoperative Continuous Infusion of Lidocaine on Analgesia in Vascular Anaesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Łukasz Krzych (Other)
Responsible Party: Sponsor-Investigator, Łukasz Krzych, Professor, Medical University of Silesia
Organization: Medical University of Silesia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCM
Record Dates: First submitted 2020-12-21; First posted 2020-12-31 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Abdominal Aorta Aneurysm; Abdominal Aorta Atheroma; Surgery; Pain, Postoperative
Keywords: lidocaine; analgesia; general anesthesia; vascular surgery; aorta
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Pain, Postoperative; Agnosia | interventions — Lidocaine; Dipyrone; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine infusion (Active Comparator): Before induction bolus of 1% lidocaine 1,5mg/kg IBW i.v., continuous infusion of 1% lidocaine intraoperatively rate 2 mg/kg IBW i.v., continuous infusion of 1% lidocaine postoperatively rate 1 mg/kg IBW i.v. for 24 hours
  Interventions: Drug: lidocaine 10mg/ml; Drug: Metamizole; Drug: Morphine
- Saline infusion (Placebo Comparator): equal volumes of placebo - 0,9% saline i.v.
  Interventions: Drug: Placebo; Drug: Metamizole; Drug: Morphine

INTERVENTIONS:
Drug: lidocaine 10mg/ml — bolus i.v. + continuous i.v. infusion
  Other Names: Lignocaine, Lidocaine
  Arms: Lidocaine infusion
Drug: Placebo — bolus i.v. + continuous i.v. infusion
  Arms: Saline infusion
Drug: Metamizole — 2,5 g i.v. BD
Drug: Morphine — continuous i.v. infusion adjusted to VAS scale score

SUMMARY:
The aim of the study is to test the effectiveness and safety of the use of lidocaine infusion in multimodal analgesic management. A group of patients undergoing vascular surgery performed with the classic technique on the aorta - with the opening of the abdominal cavity will be enrolled. The population of patients qualified for this type of vascular surgery is usually burdened with multiple diseases, mainly risk factors or cardiovascular diseases, which, combined with hemodynamic fluctuations, large fluid shifts (including bleeding) and stress for the body, affects the risk of serious cardiological complications, which in this group exceeds 5% and is the highest, according to the ESC / ESA (European Society of Cardiology / European Society of Anesthesiology) classification from 2014. Proper postoperative pain control is therefore becoming one of the key pillars of postoperative care in this group of patients.

Due to the numerous disease burden of patients and the operational specifics, the use of multimodal therapy in the management of pain is of particular importance, as the use of high doses of opioids improves hemodynamic stability, but at the same time affects the occurrence of side effects - mainly excessive sedation, respiratory disorders, hypoventilation and, consequently, for hypoxia of the heart muscle. The risk of myocardial injury in non-cardiac surgery (MINS) is significant in the light of the available literature.

Lidocaine used in intravenous infusion is one of the recommended components of multidirectional analgesia. Its adjuvant properties make it possible to reduce the amount of opioid drugs used, and thus - to reduce the frequency of their side effects. The high effectiveness of such a procedure has been proven in numerous experimental and epidemiological studies. Due to the low frequency of side effects associated with its use, the therapy has a strong recommendation for use in relieving perioperative pain. The analysis of the literature on the subject shows that there is little data assessing effectiveness of lidocaine infusion in relation to the group of patients after surgery on the abdominal aorta.

DETAILED DESCRIPTION:
All enrolled participants will be randomized, using random-number generator, to two groups - group A (intervention - perioperative continuous infusion of lidocaine) and group B (without intervention - perioperative continuous infusion of placebo). Study is designed as double-blinded: neither patients nor perioperative care givers (surgeons, anesthetists, nurses) will be aware to which group a patient has been assigned. A coordinator of randomization process will be responsible to ask an anesthetist or a nurse (a person not taking part in participant's perioperative care) to prepare a set containing respectively: 40 ml of 1% lidocaine or 40 ml of 0,9% NaCl (placebo) before surgery. Syringes will be labeled "Tested Drug". All data regarding patient's assignment to the respective groups will be available only to the coordinator of the study.

Anaesthesia will be performed by anesthetist experienced in vascular surgery. Every patient will be premedicated with midazolam (3,75mg-15 mg orally), adjusted to his/her body weight. Premedication efficacy will be assessed before induction using RASS scale (Richmond Agitation-Sedation Scale).

During induction of anaesthesia: fentanyl (0,01-0,02 mg / kg i.v.), propofol (1-2 mg/kg i.v.), atrakurium (0,5 mg/kg i.v.) will be given. Depth of anaesthesia will be monitored with BIS index (bi-spectral index) or entropy till the emergence. Patients scoring above 2 points in APFEL scale will receive antiemetic drug - ondansetron 8 mg i.v..

Intraoperative monitoring will consist of: non-invasive (NIBP) or invasive blood pressure monitoring (IBP), anesthetic agent concentration monitoring (MAC, minimal alveolar concentration), pulse oximetry (SpO2), capnometry (etCO2) and anesthetic depth monitoring as above.

During co-induction mechanical ventilation will be performed in CMV mode (controlled mechanical ventilation). Breathing frequency will be adjusted to etCO2 values. Tidal volume will be set on 6-8 ml/ kg IBW (ideal body weight) and positive end-expiratory pressure set on 5 cm H2O. Fresh gases flow mixture will be adjusted according to SpO2 92-100% values. After induction, desflurane will be used in concentrations maintaining depth of anaesthesia between 40-60 BIS/entropy values. In case of BIS/entropy values out of the range during anesthesia, all the events and duration time will be recorded. After general anesthesia mean anesthetic concentration will be counted and recorded.

All participants apart from medication used to perform general anaesthesia will receive 1g of paracetamol i.v. before induction as preemptive analgesia and intravenous bolus of the "tested drug" in the volume of 0,15 ml/kg IBW given over 1-2 minutes, followed by continuous infusion of "tested drug" with ratio of 0,2 ml/kg IBW/h intraoperatively. Postoperatively infusion will be continued with ratio 0,1ml/kg IBW/h for the next 24 hours. According to patient's assignment syringe " tested drug" will contain 1% lidocaine in group A or normal saline in group B.

Titrated doses of 0,05 mg of fentanyl i.v. will be administered as intraoperative analgesic medication. Final dose of fentanyl used during general anaesthesia will be recorded and then changed to the equivalent dose of morphine.

Blood pressure measurements will be taken every 5 minutes to assess hemodynamic stability. Initial value of patient's systolic blood pressure (SBP) and mean arterial pressure (MAP) in the operating theater will be recorded. SBP within the range from 100 to 160 mmHg and MAP >70 mmHg will be regarded as a target value (TV). In case of sudden increase in BP or HR within TV values associated with painful stimulation from operating field (assessed by experienced anesthetist), titrated dose of fentanyl will be given.

To maintain hemodynamic stability:

1. In case of decrease in BP or MAP below the TV limit: fluid challenge iv with balanced crystalloids will be commenced, especially in case of pulseoximetry or IBP wave variation. If the patient is not responding to fluid challenge, ephedrine in titrated doses of 5-10 mg will be given intravenously to maximal dose of 25 mg. If still ineffective, continues infusion of noradrenaline will be commenced.
2. In case of increase SBP above the limit: if painful response present, i.v. bolus of fentanyl in titrated doses will be given to maximal dose of 0,2 mg to achieve BP decrease to the TV. If ineffective, start re-assessment: painful stimulation present - FNT iv, no painful stimulation - urapidyl in titrated doses of 5 mg iv administered to the effect.
3. In case of increase in SBP or MAP above the limit associated with the clamping of aorta, urapidyl can be given in titrated doses as above.

Final decision regarding maintenance of hemodynamic stability in association with clinical context will be up to the anesthetist.

The number of hemodynamic interventions, BP values, total time out of the range and intraoperative fluid therapy (total amount and type of fluids, blood products), total dose of vasoactive medication will be recorded.

Postoperative care After the surgery, patients will be transferred to post surgical high-dependency unit (HDU). Proper analgesic treatment will be continued. Infusion of "tested drug" will be stopped 24 hours after the surgery.

Visual Analog Scale will be used to assess efficiency of analgesic treatment every 4 hours, with target value <4 points. Analgesia in postoperative period will consist of: continues infusion of opiate (morphine) rate adjusted according to titration method, metamizole 2,5g i.v. BD and continues infusion of "tested drug" (1% lidocaine or normal saline according to the assignment).

In case of pain exceeding 4 points in VAS scale, patient will receive bolus of 3 mg of morphine i.v., with reassessment after 15 minutes. If no improvement is obtained, second bolus of 3 mg of morphine i.v. will be administered followed by increase in the morphine infusion rate by 1 mg/h.

Any side effects in postoperative period especially associated with analgesic medication, will be recorded (according to Summary Product Characteristics, 24 hours observation), cardiovascular complications (death related to cardiovascular problems, non-fatal acute coronary syndrome; 30 days observation), incidence of post-operative delirium (POD, assessment with CAM or CAM-ICU scale, Confusion Assessment Method or Confusion Assessment Method in Intensive care Unit, 24 hour observation) Statistical analysis Statistical analysis will be performed with the use of the StatsDirect 3.1 program. The nature of the variables is verified by the Shapiro-Wilk test and the evaluation of quantile-quantile charts. Quantitative variables will be presented as arithmetic mean and standard deviation (SD) or median and interquartile range (IQR, interquartilerange). Qualitative variables are presented in the form of absolute values and percentage. The assessment of differences between the groups for quantitative variables will be performed using the Student's t-test with the variance assessment or the Mann-Whitney U test. For qualitative variables, contingency tables and a chi-square test will be used. The criterion of statistical significance is set at p˂0,05.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Vascular surgery on aorta or iliac artery
* Proximal anasthomosis of a by-pass in the abdominal cavity

Exclusion Criteria:

* Contraindications for administration of lidocaine (according to Summary Product Characteristics)
* Preoperative administration of any pain relief medication in patient, especially opioides (excluding pre-analgesia)
* Heart block second or third-degree, previous pacemaker implantation, chronic atrial fibrillation
* Antiarrhythmic medication on regular basis (excluding b-blockers prescribed due to coronary artery disease)
* Other health problems: chronic heart failure (ejection fraction LVEF<30%), epilepsy or any episode of seizure, chronic renal failure (AKIN 3-5), chronic liver failure ( class B or C in the Child-Pugh classification), Myasthenia gravis, hypoproteinemia,
* Cognitive or mental dysfunction, that prevents proper cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-07-02 (Actual)

PRIMARY OUTCOMES:
Opioid consumption in the intraoperative period | Duration of general anaesthesia
  Dose of morphine (or fentanyl changed to the equivalent dose of morphine) administered to patient to achive pain score below 4 points (VAS scale)
Opioid consumption in the postoperative period | First 24 hours after surgery
  Dose of morphine administered to patient to achive pain score below 4 points (VAS scale)
Consumption of the anesthetic agent | Duration of general anesthesia
  The Mean/median vaule of minimal alveolar concentration (MAC) necessary to maintain general anesthesia
Hemodynamic stability | Duration of general anesthesia
  Comparison of systolic and mean blood pressure value to value (5 minutes interval, comparison of exceeding 10% of the previous value, total number of exceedances)
Number of hemodynamic intervations | Duration of general anesthesia
  Total number hemodynamic interventions (total dose of vasoactive medication use according to study protocol)
Intraoperative fulid therapy | Duration of general anesthesia
  Total amount and type of fluids, blood products administered to patient

SECONDARY OUTCOMES:
The Incidence of postoperative delirium | First 72 hours (after surgery), once per shift
  Patient assessed with the CAM-ICU tool
Indicators of safety | Intraoperatively and first 24 hours (after surgery)
  Incidence of side effects (according to Summary Product Characteristics)

CONTACTS AND LOCATIONS:
Overall Officials: Łukasz J Krzych, Professor, Study Director — Medical University of Silesia, Katowice
Locations (1):
- Leszek Giec Upper-Silesia Medical Center of the Medical University of Silesia in Katowice, Katowice, Poland

REFERENCES:
- [Derived] Gajniak D, Mendrala K, Konig-Widuch G, Parzonka S, Gierek D, Krzych LJ. Effect of lidocaine on intraoperative blood pressure variability in patients undergoing major vascular surgery. BMC Anesthesiol. 2024 May 7;24(1):170. doi: 10.1186/s12871-024-02550-5. PMID 38714924